CLINICAL TRIAL: NCT01848899
Title: The Assesment of Thrombotic Markers Utilizing Ionic Versus Non-Ionic Contrast During Coronary Angiography and Intervention (AToMIC) Trial
Brief Title: Effects Contrast on Platelet Activity, Thrombosis and Fibrinolysis in Patients Undergoing Coronary Angiography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 12-02409
Record Dates: First submitted 2013-04-23; First posted 2013-05-08 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary angiography; Percutaneous coronary intervention; Contrast media; Platelet activity; Thrombin generation; Fibrinolysis
MeSH Terms: conditions — Coronary Artery Disease | interventions — iodixanol; Ioxaglic Acid; bivalirudin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ioxaglate Arm (Experimental)
  Interventions: Drug: Ioxaglate; Drug: Bivalirudin
- Iodixanol arm (Experimental)
  Interventions: Drug: Iodixanol; Drug: Bivalirudin

INTERVENTIONS:
Drug: Iodixanol — contrast media used during coronary angiography
  Other Names: Visipaque
  Arms: Iodixanol arm
Drug: Ioxaglate — contrast media used during coronary angiography
  Other Names: Hexabrix
  Arms: Ioxaglate Arm
Drug: Bivalirudin — A direct thrombin inhibitor
  Other Names: Angiomax; Angiox

SUMMARY:
The aim of this study is to determine how two different types of iodinated contrast media (CM) agents, low-osmolar ionic ioxaglate and iso-osmolar non-ionic iodixanol, affect specific markers of thrombogenesis and platelet function in patients undergoing coronary angiography, and if the use of bivalirudin, a direct thrombin inhibitor used during percutaneous coronary intervention (PCI), affects any contrast-related changes in thrombogenesis and platelet function.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be more than 18 years of age
* referred for coronary angiography and on dual anti-platelet therapy (aspirin and clopidogrel).

Exclusion Criteria:

* on warfarin
* on low molecular weight heparin within 12 hours of coronary angiography or unfractionated heparin with activated clotting time >150 at time of procedure -on cilostazol
* on persantine
* on non- steroidal anti-inflammatory medications (ibuprofen/motrin/advil, naproxen/aleve, indomethacin, sulindac, etodolac, diclofenac, celecoxib) within 72 hours of procedure
* on prasugrel (not an exclusion criteria for ST-segment elevation myocardial infarction registry
* undergoing coronary angiography via radial access
* undergoing planned diagnostic coronary angiography only
* unable to tolerate dual anti-platelet therapy
* with known allergy to CM
* received CM within 24 hours of coronary angiography
* on dialysis
* do not consent or are unable to give consent
* are participating in another competing study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Feit, MD, Principal Investigator — NYU Langone Health; Binita Shah, MD, MS, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ioxaglate Arm | Iodixanol Arm
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ioxaglate Arm | Iodixanol Arm | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 22 | 39
  >=65 years | 33 | 28 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 37 | 39 | 76

OUTCOME MEASURES:

1. Primary Outcome: Thrombin Generation Test: Baseline
Description: The thrombin generation test uses recombinant tissue factor as a stimulus to initiate thrombin generation in plasma samples. The outcome from this assay is reported as area under the curve and represents the amount of thrombin in each sample. The curve is created by measuring the generated thrombin every 20 seconds from 0 to 95 minutes post stimulus.
Time Frame: baseline
Population: A valid thrombogram was generated post-diagnostic angiography in 43/50 participants in the Ioxaglate arm and 37/50 participants in the Iodixanol arm. Thus, not all 100 participants were able to be included in analysis.
Measure: Median (Inter-Quartile Range); unit: nM*minutes
Arm/Group | Ioxaglate Arm | Iodixanol Arm
Number analyzed (Participants) | 43 | 37
nM*minutes | 1810 [1540 to 2089] | 1682 [1534 to 2147]

2. Secondary Outcome: Percent Change in Maximal Platelet Aggregation: Epinephrine
Description: Percent change in maximal platelet aggregation from pre- to post-contrast in response to 10 μM epinephrine
Time Frame: Baseline to 1 hour
Population: Sufficient volumes of blood were not available for all participants to perform the analyses required for some secondary outcomes. Thus, not all 100 participants are included in this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Ioxaglate Arm | Iodixanol Arm
Number analyzed (Participants) | 46 | 47
Percent change | 5.4 [-8.2 to 27.0] | 25.7 [.9 to 42.3]

3. Secondary Outcome: Percent Change in Maximal Platelet Aggregation: Arachidonic Acid
Description: Percent change in maximal platelet aggregation from pre- to post-contrast in response to 1600 μM arachidonic acid
Time Frame: 1 hour
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Ioxaglate Arm | Iodixanol Arm
Number analyzed (Participants) | 45 | 47
Percent change | 38.1 [10.7 to 74.3] | 36.0 [4.4 to 109.8]

4. Secondary Outcome: Percent Change in Maximal Platelet Aggregation: ADP
Description: Percent change in maximal platelet aggregation from pre- to post-contrast in response to 20 μM of ADP
Time Frame: 1 hour
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Ioxaglate Arm | Iodixanol Arm
Number analyzed (Participants) | 47 | 48
Percent change | -3 [-8.4 to 1.7] | .05 [-5.9 to 4.4]

5. Primary Outcome: Thrombin Generation Test: After Coronary Angiography
Description: as for outcome 1
Time Frame: 1 hour
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: nM*minutes
Arm/Group | Ioxaglate Arm | Iodixanol Arm
Number analyzed (Participants) | 43 | 37
nM*minutes | 649 [314 to 1347] | 681 [229 to 1237]

ADVERSE EVENTS:
Arm/Group | Ioxaglate Arm | Iodixanol Arm
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 2/50 | 1/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ioxaglate Arm (N=50) | Iodixanol Arm (N=50)
Hives/rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No